CLINICAL TRIAL: NCT00899613
Title: Study Aiming at Researching Diagnostic Markers for the Recognition of Precancerous States, Tracking, Follow-up, and the Identification of New Therapeutic Targets for Mesothelioma in Patients With Atypical Mesothelial Hyperplasia.
Brief Title: Mesothelin and Osteopontin as Diagnostic Markers in Patients With Mesothelioma or Atypical Mesothelial Hyperplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000564050; INCA-RECF0433; INCA-05-145; INCA-Mesothel
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-07

CONDITIONS: Malignant Mesothelioma; Metastatic Cancer
Keywords: localized malignant mesothelioma; lung metastases; malignant pleural effusion
MeSH Terms: conditions — Mesothelioma, Malignant; Neoplasm Metastasis; Pleural Effusion, Malignant

INTERVENTIONS:
Other: laboratory biomarker analysis
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Studying levels of mesothelin and osteopontin in samples of blood from patients with mesothelioma or atypical mesothelial hyperplasia may help doctors identify biomarkers related to cancer.

PURPOSE: This research study is looking at mesothelin and osteopontin as diagnostic markers in patients with mesothelioma or atypical hyperplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if mesothelin and osteopontin in serum can serve as early markers of malignant transformation into mesothelioma.

Secondary

* Determine if there are cytological, histological, immunohistochemical, and molecular markers of precancerous disease in tissue samples.
* Determine if SV40 has a carcinogenic role.
* Determine the relationship between the serum concentration of mesothelin and/or osteopontin and the expression of other markers and with clinical progression.

OUTLINE: This is a multicenter study.

Levels of mesothelin and osteopontin in serum (and pleural fluid, if effusion is present) are measured at baseline and 3, 6, 12, and 24 months. Patients with mesothelioma, reactional lesions, or adenocarcinoma undergo tomodensitometry (TDM) at baseline, 3, 6, and 12 months. Patients with pleural plaques only undergo TDM at 12 months.

Patients are followed for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Diagnosis of mesothelial hyperplasia and meeting 1 of the following criteria:

  * Confirmed prior exposure to asbestos and presence of pleural effusion and meets 1 of the following diagnostic criteria:

    * Mesothelioma
    * Mesothelial hyperplasia of unspecified malignancy
    * Reactional inflammatory hyperplasia
  * No asbestos exposure but pleural effusion with pleural malignant mesothelioma or pulmonary metastasis
  * Prior exposure to asbestos, no pleural effusion, and asymptomatic (pleural plaques present)
  * No prior exposure to asbestos but with benign pleural effusion
* Tissue obtained by pleuroscopy, surgical biopsy, or video-thoracoscopy available

  * Paraffin-embedded and frozen tissue available

Exclusion criteria:

* Solitary fibrous tumor
* Diffuse pleural fibrosis
* Purulent pleurisy

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Mesothelin and osteopontin concentrations in serum

SECONDARY OUTCOMES:
Cytological, histological, immunohistochemical, and molecular markers of precancerous disease in tissue samples
Role of SV40
Relationship of serum concentration of mesothelin and/or osteopontin with the expression of other markers and with clinical progression

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Galateau-Salle — University Hospital, Caen
Locations (1):
- CHU de Caen, Caen, France